CLINICAL TRIAL: NCT00398242
Title: Treatment of Stable Both-Bone Midshaft Forearm Fractures in Children: A Randomized Trial Between Treatment With Above Elbow Cast and a Combination of Above- and Below Elbow Armcast.
Brief Title: Treatment of Stable Both-Bone Midshaft Forearm Fractures in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colaris, Joost, M.D. (Individual)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Colaris03
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Last update posted 2006-11-10 (Estimated); Status verified 2006-11

CONDITIONS: Fracture; Forearm; Midshaft; Child; Treatment
Keywords: fracture; forearm; midshaft; child; treatment
MeSH Terms: conditions — Fractures, Bone | interventions — Therapeutics

INTERVENTIONS:
Device: above or below elbow cast for the last 3 weeks of treatment

SUMMARY:
We create a randomized clinical trial between the treatment with above elbow armcast alone and the treatment of above elbow in combination with a short arm cast for stable midshaft both-bone forearm fractures.

DETAILED DESCRIPTION:
children who arrive at the emergency unit with a stable both-bone midshaft forearm fracture will be asked to join the trial.

If the fracture will be stable during reposition in the operating room, a randomization between 2 kinds of plaster treatment will be done.

Outpatient clinic visits till a follow-up of 6 months. During these visits we will investigate: consolidation and dislocation on X-ray, function of both arms, complains in daily living and complications.

ELIGIBILITY:
Inclusion Criteria:

* both-bone forearm fracture
* age < 16 years
* dislocation
* stable

Exclusion Criteria:

* fracture older than 1 week
* no informed consent
* refracture
* open fracture (Gustillo 2 and 3)

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60
Dates: Start 2006-01

PRIMARY OUTCOMES:
pronation and supination

SECONDARY OUTCOMES:
complications, function, esthetics, complains in daily living, X-rays

CONTACTS AND LOCATIONS:
Overall Officials: Joost W Colaris, Drs, Principal Investigator
Locations (2):
- Netherlands (2):
  - Erasmus Medical Centre location Sophia Children's hospital, Rotterdam, South Holland
  - HAGA, location Juliana Children's Hospital, The Hague, South Holland

REFERENCES:
- [Derived] Musters L, Roth KC, Diederix LW, Edomskis PP, Benner JL, Reijman M, Eygendaal D, Colaris JW. Does Early Conversion to Below-elbow Casting for Pediatric Diaphyseal Both-bone Forearm Fractures Adversely Affect Patient-reported Outcomes and ROM? Clin Orthop Relat Res. 2024 Oct 1;482(10):1873-1881. doi: 10.1097/CORR.0000000000003100. Epub 2024 May 7. PMID 38813962